CLINICAL TRIAL: NCT06755918
Title: Effect of Video Games and Mask Painting on Anxiety and Treatment Compliance During Nebulizer Application in Children: Randomized Controlled Study
Brief Title: Video Games and Mask Painting on During Nebulizer Application in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semra Kose (Other)
Responsible Party: Sponsor-Investigator, Semra Kose, Assistant Professor (PhD, RN), Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NEU2024YLTez(1)
Record Dates: First submitted 2024-12-15; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: NEBULIZATION; Children
Keywords: Nebulizer; Child; Anxiety; Treatment Compliance; Nursing
MeSH Terms: conditions — Anxiety Disorders; Patient Compliance

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled experimental study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator)
  Interventions: Behavioral: Control
- Video game group (Experimental)
  Interventions: Behavioral: Video game
- Mask painting group (Experimental)
  Interventions: Behavioral: Mask painting

INTERVENTIONS:
Behavioral: Control — Children will be monitored when fowler is in position during the use of nebulizers. In the Fowler position, the drug will be drained into the nebulizer chamber. Mask and nebulizer connections will be completed. The patient will be told to breathe slowly and deeply. It will be examined whether sufficient steam is formed from the nebulizer device. The continuation of the application steps will be ensured until the nebulizer drug application is finished. Routine nursing care is applied during the use of nebulizer. During the use of a control group nebulizer, routine nebulizer will be used without video game and mask painting. After the receipt of the receipt, the child's anxiety scale-status scale will be requested to be filled by the child's parent and child. The treatment questionnaire developed by the researchers will be filled by the researcher. After 24 hours a day after the first nebulizer treatment of hospitalization, measurements will be made again.
  Arms: Control
Behavioral: Video game — Children will be monitoring while the fowler position during the use of nebulizers. While the Fowler position is in the position of the drug, the drug will be drained into the nebulizer reservoir. The nebul mask will be attached to cover the mouth and nose. The patient will be told to breathe slowly and deeply. It will be examined whether sufficient steam is formed from the nebulizer device. The continuation of the application steps will be ensured until the nebulizer drug application is finished. At the same time, the Water-Sorting Game will be introduced while the use of nebul will be introduced and you will be asked to play. After the receipt of the receipt, the child's anxiety scale-status scale will be requested to be filled by the child's parent and child. The treatment questionnaire developed by the researchers will be filled by the researcher. After 24 hours a day after the first nebulizer treatment of hospitalization, measurements will be made again.
  Arms: Video game group
Behavioral: Mask painting — While the Fowler position is in the position of the drug, the drug will be drained into the nebulizer reservoir. The nebul mask will be attached to cover the mouth and nose. The patient will be told to breathe slowly and deeply. It will be examined whether sufficient steam is formed from the nebulizer device. The continuation of the application steps will be ensured until the nebulizer drug application is finished. At the same time, mask painting process will be introduced while the use of nebul continues. For mask painting, six color paint will be given and the shapes and colors will be completely left to the child by leaving it to him. After the mask painting and receipt is finished, the child's anxiety scale-status scale will be requested to be filled by the child's parent and child. The treatment questionnaire developed by the researchers will be filled by the researcher. After 24 hours a day after the first nebulizer treatment of hospitalization, measurements will be made again.
  Arms: Mask painting group

SUMMARY:
The clinical features of respiratory system diseases seen in childhood are generally moderate and improve in a short time. Respiratory system diseases are divided into two as upper respiratory system diseases and lower respiratory system diseases. The respiratory tract, from the mouth and nose, which are the upper respiratory tract, to the glottis (nasal mucosa, nasopharynx, oropharynx, sinuses, middle ear tonsils and epiglottis) and the infections that occur in these sections are called upper respiratory tract infections (URTI). Lower respiratory system diseases are considered as tuberculosis, asthma, cystic fibrosis and bronchopulmonary dysplasia. The most common diseases in children are respiratory tract diseases. The diseases that are considered as priorities for each age group vary. According to the Turkish Thoracic Society, the incidence of lower respiratory tract infections (LRTI) between the ages of 0-5 is 29%. According to TUIK 2022 data, upper respiratory tract infections are the most common infectious diseases experienced by children between the ages of 0-6 with a rate of 31.3%, and lower respiratory tract infections are the third with a rate of 6.9%. In children between the ages of 7-14, upper respiratory tract infections are the most common with a rate of 27.1%, and lower respiratory tract infections are the third with a rate of 5.3%.

DETAILED DESCRIPTION:
The treatment of respiratory system diseases includes maintaining airway patency, using antibiotics and corticosteroids, and oxygen support. The most preferred is bronchodilator - vasoconstriction and bronchodilation (nebule therapy). Nebulizer use reduces symptoms by reducing wheezing, shortness of breath, and edema in the respiratory tract, and therapeutics (saline fluids, bronchodilators, epinephrine, anticholinergic agents, and corticosteroids) used are used as a treatment option. The use of nebulizer drugs is used as an emergency treatment method in both children and adults, especially in respiratory system diseases, all over the world and in Turkey. In addition, their use in the treatment of lung diseases is increasing. The main purpose of inhalation treatment is to send smaller amounts of medication directly to the respiratory tract as soon as possible, to deliver drug particles to the farthest lobes of the lungs, to eliminate airway stenosis in the respiratory system and to regulate the amount of mucus.

In children, the process of hospitalization, treatment, and the devices used can be traumatic. Many devices used in the hospital, such as the use of nebulizers, the sounds of the devices, unfamiliar people, unfamiliar environments, dependence on caregivers, unfamiliar tools and equipment, traumatic and painful invasive procedures, separation from family and friends, disruption of routines such as sleep, eating, playing, and school can affect children's anxiety levels and compliance with treatment. The pain and suffering they experience during procedures can be reduced by using distraction methods. One of the distraction methods is therapeutic play. Therapeutic play should be used as an effective method to minimize the negative effects of procedures and to support the child in developing effective coping methods. It has been observed in literature studies that children who use nebulizers together with therapeutic play have decreased fear, pain, anxiety and stress levels. In the study conducted by Kırkan et al. (2023), it was observed that nebulizer treatment with a toy nebulizer and a toy mask decreased children's anxiety levels. In another study conducted by Kurtuncu et al. (2019), it was observed that 3-dimensional nebulizer treatment reduced psychosocial symptoms seen in children. In another study, it was determined that education given with a toy-type nebulizer reduced anxiety levels in children. Therapeutic play allows effective cooperation with the child by understanding the child's behavior. Therapeutic play has an important measure in ensuring that children comply with treatment, display positive behavior, and improve care. This study, which can be easily applied by nurses in the hospital environment before, during, and after medical, invasive procedures, will also ensure children's compliance with treatment and is thought to contribute to the literature; will be conducted to examine the effects of video games and mask painting on anxiety and treatment compliance during nebulizer application in children.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 7-12
* Receiving the first nebulization treatment after hospitalization
* Able to speak and read Turkish
* Receiving nebulizer treatment
* Children who agree to participate in the study and children whose parents agree to participate in the study

Exclusion Criteria:

* Those who are allergic to paint
* Those who have a chronic disease and routinely use a nebulizer
* Those who are connected to any respiratory device (mechanical, etc.)
* Those who did not complete the intervention and wish to withdraw from the study
* Those who have any body function deficiency that prevents coloring or tablet games

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | The introductory information form will be filled out by the researcher during the first nebule treatment of the children's hospitalization. (Approximately 5 minute)
  It was created by the researcher in line with the literature in order to obtain the child's sociodemographic and disease information. The form contains nineteen questions including the child's age, gender, school attendance status, previous nebulizer use status and the reaction if the child has previous nebulizer use experience.
Child Anxiety Scale-State | After the nebulization process is completed, the child anxiety scale-state scale will be asked to be filled out by the child's parent and the child. (Approximately 10minute). Repeat measurements will be taken 24 hours after the first nebulizer treatment.
  Child Anxiety Scale-State was developed by Ersıg and his colleagues in 2013 to measure the state anxiety of children between the ages of 4-10, and its validity and reliability in our country were determined by Ozalp Gerceker and his colleagues (2018). The child anxiety scale looks like a thermometer with 10 sections and is very easy to use. It indicates that anxiety increases as you go from bottom to top (0=calm, 10=very anxious). The child is asked to mark the sections on the scale that they feel 'right now'. In the literature research, it was seen that the scale was used between the ages of 7-12.
Treatment Adherence Questionnaire | The treatment compliance questionnaire developed by the researchers will be filled out by the researcher. (Approximately 5 minute) Repeat measurements will be taken 24 hours after the first nebulizer treatment.
  The form created by the researchers in line with the literature is a form created to measure children's compliance during treatment. It includes children's reactions and vital signs. This form will be sent to academicians and specialist nurses who are experts in the field of child health and disease nursing and will be presented for expert opinion. The form, which has been finalized and the expert opinion has been completed, will be applied to children during and after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No